CLINICAL TRIAL: NCT04755569
Title: Clinical Investigation of the ODOCOR II CCM™ Leads in Patients With Optimizer System Implant
Brief Title: Optimizer System With ODOCOR II CCM™ Leads
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: Impulse Dynamics
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Evaluate the Safety and Useability of the ODOCOR II Intra-cardiac Lead

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ODOCOR II CCM LEADS — ODOCOR II CCM LEADS Implantation

SUMMARY:
The objective of the ODOCOR II CCM lead study is to evaluate the safety and useability of the ODOCOR II intra-cardiac lead specifically intended to deliver CCM as an accessory lead to the Optimizer IPG.

DETAILED DESCRIPTION:
Design A prospective, multi-center, single arm open label study, 12-month study of 400 ODOCOR II CCM™ leads in 200 subjects .

Method Subjects shall be enrolled that have been diagnosed with NYHA Class III-IV heart failure and left ventricular ejection fraction (25-45% inclusive). Eligible subjects will receive the Optimizer IPG device implant with 2 ODOCOR II CCM leads. Subjects will return for follow-up visits at 2-weeks, 6 months and 12 months following the device implant.

Endpoints Primary Safety endpoint

The primary safety endpoint is the incidence of lead-related complication free rate at 12 months post-index implantation procedure compared to the incidence previously described in the literature for pacing therapy leads.

Secondary Safety endpoint

The secondary safety endpoint is an assessment of the lead-related "observations" occurring during the 12-month study.

Primary Efficacy endpoint The total amount of CCM delivered to the cardiac tissue of the right ventricle (measured by CCM percentage) will be measured over a period of 12 months.

Secondary Efficacy endpoint Change in QOL, as measured by the Minnesota Living with Heart Failure Questionnaire (MLWHFQ), from baseline to 12 months following index implantation procedure.

Additional Endpoints Handling characteristics of the lead will be evaluated by the implanting physician. Ease of insertion, lead visibility on x-ray, and the ability to visualize the helix deployment will be assessed via a questionnaire administered at the completion of an implant procedure.

Patients, sites Four hundred (400) ODOCOR II CCM leads will be implanted in 200 eligible subjects from up to 40 sites in Europe.

Duration The total investigation is expected to last approximately 3 years , including enrollment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Patient signed and dated informed consent form
2. Male or non-pregnant female, aged 18 or older
3. Left ventricular ejection fraction of 25-45% (inclusive)
4. Diagnosed with NYHA Class III or IV heart failure
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Medically stable and with no significant mental illness in the judgement of the principal investigator

Exclusion Criteria:

1. Infiltrative or inflammatory cardiomyopathy (e.g. amyloid, hemochromatosis, myocarditis, hypertrophic cardiomyopathy, Fabry's disease, cardiac tumor)
2. Primary heart failure due to uncorrected mitral valve disease, or mitral valve repair or clip within 3 months of the baseline testing visit.
3. IV inotropes, hemofiltration, or any form of positive inotropic support within 30 days before the baseline testing visit, including continuous IV inotrope therapy
4. Myocardial infarction within 3 months of the baseline testing visit.
5. Undergone a CABG procedure within 3 months90 days or a PTCA procedure within 30 days of the baseline testing visit.
6. Undergone a cardiac ablation procedure within 90 days prior to consent.
7. Prior heart transplant or ventricular assist device
8. Mechanical tricuspid valve
9. Receiving cardiac resynchronization therapy (CRT) or indicated for Class I CRT implantation according to the ACCF/AHA/HRS guidelines for device-based therapy
10. Currently on dialysis
11. Currently undergoing active chemotherapeutic and/or radiation treatment for cancer
12. Participating in another cardiac investigational device study at the same time
13. Patient is in a vulnerable population (such as significant mental disability, prisoner) that in the judgement of the PI impedes ability to provide informed content.
14. Expected lifespan of less than 12 months from time the baseline testing visit.
15. Resting heart rate >110 bpm at the time of the baseline testing visit
16. Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
17. Subjects currently admitted to the hospital with a primary diagnosis of heart failure

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total investigation is expected to last approximately 3 years , including enrollment and follow-up periods.
  Four hundred (400) ODOCOR II CCM leads will be implanted in 200 eligible subjects from up to 40 sites in Europe
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety endpoint | 12 months
  The primary safety endpoint is the incidence of lead-related complication free rate at 12 months post-index implantation procedure compared to the incidence previously described in the literature for pacing therapy leads.
Primary Efficacy endpoint | 12 month
  The total amount of CCM delivered to the cardiac tissue of the right ventricle (measured by CCM percentage) will be measured over a period of 12 months.

SECONDARY OUTCOMES:
Secondary Safety endpoint | 12 month
  The secondary safety endpoint is an assessment of the lead-related "observations" occurring during the 12-month study.
Secondary Efficacy endpoint | 12 month
  Change in QOL, as measured by the Minnesota Living with Heart Failure Questionnaire (MLWHFQ), from baseline to 12 months following index implantation procedure.

OTHER OUTCOMES:
Additional Endpoints | at implant
  Handling characteristics of the lead will be evaluated by the implanting physician. Ease of insertion, lead visibility on x-ray, and the ability to visualize the helix deployment will be assessed via a questionnaire administered at the completion of an implant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano DeVivo, MD, Principal Investigator — Monaldi Hospital
Locations (40):
- Germany (20):
  - Klinik am Plattenwald, Heilbronn, Baden-Wurttemberg
  - St. Anna Krankenhaus, Sulzbach-Rosenberg, Bavaria
  - St. Josefs-Hospital Wiesbaden GmbH, Wiesbaden, Hesse
  - Elbe Klinikum Stade, Stade, Lower Saxony
  - Augusta-Kranken-Anstalt Bochum-Mitte, Bochum, North Rhine-Westphalia
  - Krankenhaus Marie-Hilf Stadtlohn, Stadtlohn, North Rhine-Westphalia
  - Herzzentrum Dresden, Dresden, Saxony
  - Klinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - DRK Kliniken Berlin Koepenick, Berlin
  - Charité Berlin Campus Virchow, Berlin
  - Evangelisches Klinikum Bethel, Bielefeld
  - Regiomed Kliniken-Coburg, Coburg
  - SRH Krankenhaus Waltershausen-Friedrichroda, Friedrichroda
  - Marienhospital, Gelsenkirchen
  - Asklepios Klinik St. Georg, Hamburg
  - Schoen Klinik Hamburg Eilbek, Hamburg
  - Evangelisches Krankenhaus Herne, Herne
  - St. Marien-Hospital Klinikum Luenen, Lünen
  - Universitaetsklinikum UMM, Mannheim
  - Niels-Stensen-Kliniken Marienhospital Osnabrück GmbH, Osnabrück
- Italy (15):
  - Azienda Ospedaliera Dei Colli-Monaldi, Naples, Campania
  - Ospedale "Sacra Famiglia" - Fatebenefratelli dell', Erba, Lombardo Veneta
  - Ente Ecclesiastico Ospedale Generale Regionale "F.Miulli" Cardiologia e U.T.I.C., Acquaviva delle Fonti
  - Ospedale C. e G. "Mazzoni", Ascoli Piceno
  - Ospedale San Paolo, UOC Cardiologia ed UTIC, Bari
  - Azienda Ospedaliero Universitaria Consorziale - Policlinico di Bari U.O.C Cardiologia Ospedaliera, Bari
  - IRCCS Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Azienda Sanitaria Provinciale di Cosenza "Ospedale di Castrovillari, Castrovillari
  - ASL TO 4 - Presidio Ospedaliero Riunito sede di Cirie, Cirié
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Maggiore della Carita, Novara
  - Gruppo Synergo - Casa Di Cura Pierangeli, Pescara
  - Presidio Ospedaliero Sant'Andrea, Vercelli
  - Ospedale San Bortolo di Vicenza - Azienda UlSS 8 Berica, Vicenza
- Spain (5):
  - Complejo Hospitario Torrecardenas, Almería
  - Hospital Virgen de las Nieves, Granada
  - Hospital 12 de Octubre, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Clinico U. de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No